CLINICAL TRIAL: NCT00330512
Title: Maternal Hypotension During Elective Cesarean Section and Short Term Neonatal Outcome.
Brief Title: Maternal Hypotension During Cesarean Section and Short Term Neonatal Outcome.
Status: Terminated | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Ayala Maayan, Sehba Medical Center
Other Study IDs: SHEBA-06-4117-AM-CTIL
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Elective Cesarean Section; Maternal Hypotention
Keywords: regional anestesia; cesarean section; hypotention; newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
About 20-25% of deliveries are by cesarean section. Most are elective with use of regional anesthesia (spinal/epidural). Drop of blood pressure after regional anesthesia is common. It have the risk of reduction of blood flow to the placenta and the fetus.

No studies had followed the newborns their first days of live,of mothers who developed hypotension in durins CS.

DETAILED DESCRIPTION:
A reterospective study of all full term babies, born in elective cesarean section with use of regional anesthesia. Two groups will be define rgarding maternal hypotention following regional anesthesia - maternal hypotention (study group) or normal maternal BP. The definition of Maternal hypotension: decrease in 10% or more in mean BP in compared to first BP taken at admition.

Data will colect from mothers and neonates records as well as operation data. Maternal data: gravida, parity, diseases, medications, demographics, and all data regarding the operation (blood pressures, Heart rates, saturation, treatment given etc.).

Infant data: gestational age, birth weight, sex, Apgar, cord pH, clinical manifestations, medications, time of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* fullterm infants, born by elective cesarean section using regional anasthesia.

Exclusion Criteria:

* preterms, urgent CS, CS using general anasthesia, Multiple pregnancy, Congenital malformations.

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayala Maayan, MD, Principal Investigator — Sheba Medical Center